CLINICAL TRIAL: NCT00592280
Title: Two-Layer Method Preservation and Resuscitation of the Cadaveric Pancreas Before Transplantation
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Logistic problems with adequately timely organ collection and transport
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0047-07-FB
Record Dates: First submitted 2007-12-17; First posted 2008-01-14 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Graft Pancreatitis
Keywords: Pancreas transplantation; graft pancreatitis; Two-layer method; organ preservation
MeSH Terms: conditions — Pancreatitis, Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pancreas Preservation (Experimental): The pancreas will be preserved before transplantation in an oxygenated system containing highly oxygenated liquid perfluorocarbon (perfluorodecalin, C10F18. The perfluorocarbon combines low toxicity with a capacity to dissolve 75 times more oxygen than the UW solution used in standard pancreas storage. When preserved under these conditions, the pancreas absorbs oxygen by diffusion and steadily consumes it, supporting sufficient aerobic metabolism to maintain tissue ATP concentrations at near-physiologic levels and prevent, or even reverse, pancreas anoxic injury.
  Interventions: Drug: Two-Layer Method pancreas preservation system drug; Device: Two-Layer Method pancreas preservation system device

INTERVENTIONS:
Drug: Two-Layer Method pancreas preservation system drug — Preserving the pancreas before transplantation in an oxygenated system containing highly oxygenated liquid perfluorocarbon (perfluorodecalin, C10F18. The perfluorocarbon combines low toxicity with a capacity to dissolve 75 times more oxygen than the UW solution used in standard pancreas storage. When preserved under these conditions, the pancreas absorbs oxygen by diffusion and steadily consumes it, supporting sufficient aerobic metabolism to maintain tissue ATP concentrations at near-physiologic levels and prevent, or even reverse, pancreas anoxic injury.
  Other Names: pancreas preservation
Device: Two-Layer Method pancreas preservation system device — Preserving the pancreas before transplantation in an oxygenated system containing highly oxygenated liquid perfluorocarbon (perfluorodecalin, C10F18. The perfluorocarbon combines low toxicity with a capacity to dissolve 75 times more oxygen than the UW solution used in standard pancreas storage. When preserved under these conditions, the pancreas absorbs oxygen by diffusion and steadily consumes it, supporting sufficient aerobic metabolism to maintain tissue ATP concentrations at near-physiologic levels and prevent, or even reverse, pancreas anoxic injury.
  Other Names: pancreas preservation

SUMMARY:
The purpose of this project is to compare the effect of oxygenated preservation of the pancreas before transplantation using the "Two-Layer Method" (TLM) against outcomes previously experienced with organs preserved using only standard University of Wisconsin (UW) storage solution. It is our hypothesis that TLM preservation will reduce the frequency and severity of complications of pancreas transplantation, increase the number of organs acceptable for transplantation, and spare individual patients and their families suffering and hardship.

DETAILED DESCRIPTION:
Two-Layer Method (TLM) preservation consists of a storage chamber containing a layer of highly oxygenated, water-immiscible liquid perfluorocarbon (perfluorodecalin, C10F18) surmounted by a layer of conventional UW (or similar) organ preservation solution. The perfluorocarbon is sufficiently dense (~2 g/ml) that the pancreas floats on top of it, in contact with both layers. The perfluorocarbon combines low toxicity with an oxygen content 75 times greater than the UW solution used in standard pancreas storage. When preserved under these conditions, the pancreas absorbs oxygen by diffusion and steadily consumes it, supporting sufficient aerobic metabolism to maintain tissue ATP concentrations at near-physiologic levels and prevent, or even reverse, pancreas anoxic injury. In animal models of pancreas ischemic and storage injury, TLM preservation has been strikingly successful at improving the outcome of both islet isolation and pancreas transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Listed for pancreas transplantation at the University of Nebraska Medical Center

Exclusion Criteria:

* Ineligibility for medical/surgical/psychosocial reasons for listing for pancreas transplantation at the University of Nebraska Medical Center.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Post-transplantation adverse event frequency | 1 year
  Post-transplantation adverse event frequency (graft thrombosis, hemorrhage, peri-pancreatic abscess, re-laparotomy, cadaver duodenum leak, pseudo-aneurysm formation, rejection, graft failure, patient death)

SECONDARY OUTCOMES:
Standard post-transplantation morbidity endpoints | 1 year
  Standard post-transplantation morbidity endpoints including fungal, bacterial, and viral infections, and incidence and rate of stroke and heart attack. Length of hospital stay and re-admission and re-operation rates will also be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: R Brian Stevens, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- The Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Matsumoto S, Kandaswamy R, Sutherland DE, Hassoun AA, Hiraoka K, Sageshima J, Shibata S, Tanioka Y, Kuroda Y. Clinical application of the two-layer (University of Wisconsin solution/perfluorochemical plus O2) method of pancreas preservation before transplantation. Transplantation. 2000 Sep 15;70(5):771-4. doi: 10.1097/00007890-200009150-00010. PMID 11003355
- [Background] Hiraoka K, Kuroda Y, Suzuki Y, Fujino Y, Tanioka Y, Matsumoto S, Sakai T, Kandaswamy R, Sutherland DE. Outcomes in clinical pancreas transplantation with the two-layer cold storage method versus simple storage in University of Wisconsin solution. Transplant Proc. 2002 Nov;34(7):2688-9. doi: 10.1016/s0041-1345(02)03376-6. No abstract available. PMID 12431575